CLINICAL TRIAL: NCT04449133
Title: Crossover, Double-blind, Phase 2 Study of AD128 Versus Placebo in Obstructive Sleep Apnea
Brief Title: Study of AD128 Versus Placebo in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: YGHEA, CRO Division of Ecol Studio spa (Industry); STM Pharma PRO srl (Unknown); Apnimed Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-004917-15
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Apnea Hypopnea Index
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Patients who meet the eligibility criteria will be assigned alternatively to the the treatment with a AD128 or matching placebo. After 7 days of treatment and a washout period, the patients will crossover to the other arm for 7 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group 1 (Experimental): AD128 for 7 days, then, after a wash-out period of 7-10 days, placebo for 7 days
  Interventions: Drug: AD128; Drug: Placebo
- Treatment Group 2 (Experimental): Placebo for 7 days, then, after a wash-out period of 7-10 days, AD128 for 7 days
  Interventions: Drug: AD128; Drug: Placebo

INTERVENTIONS:
Drug: AD128 — Oral administration of two capsules before sleep for 7 days.
Drug: Placebo — Oral administration of two capsules before sleep for 7 days.

SUMMARY:
Obstructive Sleep Apnea (OSA) is the most common and serious of the sleep disorders. Long-term, OSA is associated with increased morbidity and mortality, with a number of adverse cardiovascular, neurocognitive, metabolic, and daytime functioning consequences. No drugs are currently approved for OSA treatment.

This is a randomized, double blind, placebo controlled, cross-over, inpatient phase 2 clinical trial to examine the efficacy and the safety of a fixed dose level of AD128 in patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to understand the nature of the study and to give free informed consent
* AHI ≥ 15 on screening/baseline PSG
* Any of the following conditions should be met:

  1. Documented prior PSG within 1 year demonstrating AHI of 15 or higher
  2. Documented Continuous Positive Airway Pressure (CPAP) intolerance or poor compliance (compliance is defined as self-reported use of CPAP 4 hours per night for 70% of nights) or CPAP-naïve.
  3. Patients who have been using CPAP at least 4 hours nightly for at least 70% of the nights are eligible only if CPAP is not used for 2 weeks prior to the screening/study baseline PSG.
* Epworth Sleepiness Scale (ESS) score ≥ 4 for patients not using CPAP
* Previous surgical treatment for OSA is allowed if ≥ 1 year prior to enrollment.
* BMI between 18.5 and 40.0 kg/m2, inclusive

Exclusion Criteria:

* History of narcolepsy.
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease or hypertension requiring more than 3 medications for control.
* Clinically significant neurological disorder, including epilepsy/convulsions
* History of schizophrenia, schizoaffective disorder or bipolar disorder according to - Diagnostic and Statistical Manual of Mental Disorders-V (DSM V) or International Classification of Disease X edition criteria.
* History of attempted suicide or suicidal ideation within 1 year prior to screening, or current suicidal ideation.
* Positive history for abuse of drugs or substance use disorder as defined in DSM-V within 12 months prior to Screening Visit.
* A significant illness or infection requiring medical treatment in the past 30 days.
* Clinically significant cognitive dysfunction.
* Untreated narrow angle glaucoma.
* Women who are pregnant or nursing.
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.
* History of using devices to affect participant sleeping position for the treatment of OSA, e.g. to discourage supine sleeping position, may enroll as long as the devices are not used during participation in the study.
* History of oxygen therapy.
* Use of medications from the list of disallowed concomitant medications.
* Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, or monoamine oxidase inhibitors (MAOI) or linezolid within 14 days of the start of treatment, or concomitant with treatment.
* Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.
* Central apnea index > 5/hour on baseline PSG
* Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.
* Patients considered by the investigator, for any reason, unsuitable candidates to receive AD128 treatment or unable or unlikely to understand or comply with the dosing schedule or study evaluations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea Index (AHI) | From the screening/baseline to the last day of treatment (7 days after the start of each treatment period).
  The percentage change of mean AHI will be compared between treatment groups.

SECONDARY OUTCOMES:
AHI decrease ≥50% | From screening/baseline to the last day of treatment (7 days after the start of each treatment period).
  The proportion of patients with AHI decrease ≥50% will be calculated.
AHI<15/hour | From screening/baseline to the last day of treatment (7 days after the start of each treatment period).
  The number of patients with AHI <15/hour measured during the inpatient night Polysomnography will be compared between treatment groups.
Change in Epworth Sleepiness Scale (ESS) | From screening/baseline to the last day of treatment (7 days after the start of each treatment period).
  The ESS is a self-administered questionnaire which measures the daytime sleepiness. The ESS score can range from 0 to 24. The change will be measured in terms of difference from baseline and between treatment groups.
Change in Karolinska Sleepiness Scale (KSS) | From screening/baseline to the last day of treatment (7 days after the start of each treatment period).
  The KSS is a self-reported 9-points scale which measure the subjective level of sleepiness at a particular time during the day. The change will be measured in terms of difference from baseline and between treatment groups.
Patient Global Impression of OSA Severity (PGI-S) | From screening/baseline to the last day of treatment (7 days after the start of each treatment period).
  The PGI-S is a single question asking the patient to rate on a scale, ranging from 0 to 4, the severity of the OSA condition at that time.
Change in Psychomotor Vigilance Test (PVT) | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
  PVT is a chronometric measure of a patient's reaction time to a visual stimulus. PVT reaction times/lapses and failures to react will be measured. The change will be measured in terms of difference from baseline and between treatment groups.
Change in Oxygen Desaturation Index (ODI) 3% | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
  The number of times per hour of sleep that the blood's oxygen level drops by 3% from baseline will be measured by means of a CE marked oximeter capable of nightly recording and storage of data for the entire at-home period. The change in mean value from baseline will be compared between treatment groups.
Change in total time with Oxygen Saturation (SaO2) <90% | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
Change in mean SaO2 | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
Change in minimum SaO2 | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
Change in arousal index | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
  The number of arousals will be registered during the polysomnography and reported as a frequency per hour of sleep. The change in mean value from baseline will be compared between treatment groups.
Change in periodic limb movement | From screening/baseline to last day of treatment (7 days after the start of each treatment period).
  The number of periodic limb movements will be measured during the polysomnography. The change in mean value from baseline will be compared between treatment groups.
Oxygen Desaturation Index 4% | For the entire at home treatment period: days 1-7 (before crossover) and days 15-20 (after crossover)
  The number of times per hour of sleep that the blood's oxygen level drops by 4% or more from baseline will be measured by means of a CE marked oximeter capable of nightly recording and storage of data. The average numbers will be compared between treatment groups.
Adverse Events (AE) | From screening/baseline to 4 weeks after last day of treatment.
  All adverse events occurring to patients after recruitment in the study will be recorded. The total number of AEs, their severity and their seriousness will be compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Perger, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano,Ospedale San Luca, Milan, Italy

REFERENCES:
- [Derived] Perger E, Taranto Montemurro L, Rosa D, Vicini S, Marconi M, Zanotti L, Meriggi P, Azarbarzin A, Sands SA, Wellman A, Lombardi C, Parati G. Reboxetine Plus Oxybutynin for OSA Treatment: A 1-Week, Randomized, Placebo-Controlled, Double-Blind Crossover Trial. Chest. 2022 Jan;161(1):237-247. doi: 10.1016/j.chest.2021.08.080. Epub 2021 Sep 20. PMID 34543665